CLINICAL TRIAL: NCT04262349
Title: The Effect of the Training Program on Sleep Quality
Brief Title: The Effect of the Training Program on Increasing Sleep Quality in Pregnancy to Maternal Sleep Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Habibe BAY, research assistant, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0000-0001-5786-4385
Record Dates: First submitted 2020-02-05; First posted 2020-02-10 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Intervention Model Description: : The study was a randomized controlled training intervention study. Sample size was calculated with G * Power 3.0.10 program with an effect size of 0.3 (medium effect level) and a power of 80%. A total of 180 pregnant women were identified as 90 in the intervention group and 90 in the control group. Considering that data will be lost due to reasons such as discontinuation and exclusion criteria during pregnancy 10% more of the determined number was included in the study and the sample size was calculated as 198 pregnant women and 252 pregnant women were reached during the study. 36 pregnant women in the intervention group and 35 pregnant women in the control group were excluded from the study for different reasons and the study was completed with 181 pregnant women (90: control: 91). The groups were determined by randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): Every week because of differences in the number of pregnant women who attended the school participating women were divided into two groups using a random number table created in the program via the computer itself. The purpose of the study was explained to pregnant women, informed consent form and data collection tools of the study were collected by face to face interview technique. In the first interview to all pregnant women; Personal Information Form, Course Information Form, Pittshburg Sleep Quality Index (PUKI) and General Self-Efficacy Scale were applied. Pregnant women in the intervention group were given a two-session training program to improve sleep quality and "Sleep Guide" and "Safe Baby Sleep Conditions Brochure".
  Interventions: Behavioral: sleep education
- control (No Intervention): Pregnant women in the control group were subjected to routine practice without any training given by the researcher. Four weeks after the completion of the sleep training, all pregnant women were contacted by telephone and the data collection tools were applied for the second time and the final test applications were completed. After completion of the data collection process made a new plan for training to improve the quality of sleep to pregnant women in the control group and the "Sleep Guide" and "Safe Baby Sleep Conditions Brochure" is given.

INTERVENTIONS:
Behavioral: sleep education — As a training program to increase sleep, pregnant women will be given 2 training sessions per week for two weeks and four sessions in total for 60 minutes.
  Arms: intervention

SUMMARY:
The aim of this study is to compare the control group and the intervention to be applied to the education program used to increase sleep quality in nulliparous women.

DETAILED DESCRIPTION:
The study was a randomized controlled training intervention study in the pre-test and post-test order. The population of the study consisted of nulliparous pregnant women who applied to the Konya Dr. Ali Kemal Belviranlı Maternity and Children Hospital Pregnancy School and met the criteria for inclusion in the study at time of the study. Sample size was calculated with G * Power 3.0.10 program with an effect size of 0.3 (medium effect level) and a power of 80%. A total of 180 pregnant women were identified as 90 in the intervention group and 90 in the control group. Considering that data will be lost due to reasons such as discontinuation and exclusion criteria during pregnancy 10% more of the determined number was included in the study and the sample size was calculated as 198 pregnant women and 252 pregnant women were reached during the study. 36 pregnant women in the intervention group and 35 pregnant women in the control group were excluded from the study for different reasons and the study was completed with 181 pregnant women (90: control: 91). The groups were determined by randomization. During the conduct of the study, all pregnant women who applied to the pregnant school and met the criteria for participation in the study were recorded in the pre-training registry and numbered in the order of registration. Every week because of differences in the number of pregnant women who attended the school participating women were divided into two groups using a random number table created in the program via the computer itself. The purpose of the study was explained to pregnant women, informed consent form and data collection tools of the study were collected by face to face interview technique. In the first interview to all pregnant women; Personal Information Form, Course Information Form, Pittshburg Sleep Quality Index (PUKI) and General Self-Efficacy Scale were applied. Pregnant women in the intervention group were given a two-session training program to improve sleep quality and "Sleep Guide" and "Safe Baby Sleep Conditions Brochure". Pregnant women in the control group were subjected to routine practice without any training given by the researcher. Four weeks after the completion of the sleep training, all pregnant women were contacted by telephone and the data collection tools were applied for the second time and the final test applications were completed. After completion of the data collection process made a new plan for training to improve the quality of sleep to pregnant women in the control group and the "Sleep Guide" and "Safe Baby Sleep Conditions Brochure" is given.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women
* between 28 and 32 gestational weeks

Exclusion Criteria:

* under 18 years old

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2018-12-30 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Sleep Quality | change in sleep quality in the 4th week of education
  Pittshburg Sleep Quality Index (PUKI):
  PUKI is a self-report scale that evaluates sleep quality and disorders in the past month.
  It consists of 24 questions in total, 19 of which are self-report based questions.
  The last 5 questions are not included in the scoring, they are used for clinical evaluation.
  Each item of the scale is evaluated as 0-3 points.
  Seven "component" scores are created from nineteen items. While some components consist of evaluating a single substance, some components are the result of combining several items.
  Components that make up the scale; subjective sleep quality, sleep delay, sleep duration, habitual sleep effectiveness, sleep disorders, use of sleeping pills and daytime dysfunction.
  The scale total score is obtained by calculating the points of these seven components and the maximum scale score that can be obtained is 21.
  Increased score indicates poor sleep quality.
  A total scale score of 5 and above is expressed as bad sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Neriman Soğukpınar, Study Director — Ege University
Locations (1):
- Ege University, Selçuk, Eyalet/Yerleşke, Turkey (Türkiye)

REFERENCES:
- [Derived] Bay Ozcalik H, Sogukpinar N. The Effect of Sleep Enhancement Educational Program on Maternal Sleep Quality for Nulliparous Pregnant Women: A Randomized-Controlled Trial. Int J Behav Med. 2025 Feb;32(1):11-20. doi: 10.1007/s12529-024-10261-x. Epub 2024 Jan 29. PMID 38286916